CLINICAL TRIAL: NCT02267668
Title: Subsymptom Threshold Exercise Protocol (STEP) to Recovery Following Mild Traumatic Brain Injury: A Pilot Randomized Controlled Clinical Trial
Brief Title: Subsymptom Threshold Exercise Protocol Following Mild TBI
Acronym: STEP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospitals Cleveland Medical Center (Other)
Responsible Party: Principal Investigator, Christopher M. Bailey, Neuropsychologist and Director of Concussion Program, Neurological Institute, University Hospitals Cleveland Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 11-13-04
Record Dates: First submitted 2014-10-14; First posted 2014-10-17 (Estimated); Last update posted 2018-05-14 (Actual); Status verified 2018-05

CONDITIONS: Traumatic Brain Injury
Keywords: concussion; sports concussion; exercise therapy
MeSH Terms: conditions — Brain Injuries, Traumatic; Brain Concussion

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- STEP arm (Experimental): The Baseline Evaluation Session will include formal neuropsychological evaluation, postural stability evaluation, and an education session (education about mTBI, mTBI recovery, and expected outcomes from mTBI).
  Intervention includes exercise tolerance evaluations, 3 times per week exercise by physical therapist. Self report of symptoms and exertion.
  Interventions: Behavioral: STEP
- Control (Active Comparator): The Baseline Evaluation Session will include formal neuropsychological evaluation, posturalstability evaluation, and an education session (education about mTBI, mTBI recovery, and expected outcomes from mTBI).
  Control protocol includes instructions for stretching, instructions for restricting physically demanding activity during first 3 weeks of study; instructions for light, self-guided daily exercise in last 3 weeks of study. Self report of symptoms and exertion.
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: STEP — Physical therapists guide participants through novel set of assigned exercises
  Other Names: Subsymptom Threshold Exercise Protocol
  Arms: STEP arm
Behavioral: Control — Participants self-guide through standard exercises
  Arms: Control

SUMMARY:
The study will monitor outcomes of two interventions to develop a best practice in the treatment of mild Traumatic Brain Injury (mTBI).

DETAILED DESCRIPTION:
The proposed pilot randomized controlled clinical trial (RCCT) will provide preliminary data to examine the effect of a novel intervention to promote brain health after mild Traumatic Brain Injury (mTBI). The study will implement a randomized controlled clinical trial of a 6 week exercise intervention (STEP) for participants with persistent mTBI symptoms, comparing STEP to standard of care practice in the controls. We will demonstrate the feasibility and acceptability of the STEP intervention. We hypothesize that STEP will lead to meaningful improvement on objective measures of self-reported mTBI symptoms, formal neuropsychological performance, and postural stability.

ELIGIBILITY:
Inclusion Criteria:

1. Participants who have sustained a concussion and have not experienced symptom resolution by 4 weeks, as indicated by a Post-Concussive Scale - Revised (PCS-R) score of 20 or higher at 4 weeks post-injury or beyond;
2. Participants are high school and college age (14-22 years old);
3. English speaking. -

Exclusion Criteria:

1. Outside of age range for the study (High school or college age)
2. Have physical injuries or comorbidities that restrict the athlete from engaging in the exercise intervention
3. Not fluent in English -

Ages: 14 Years to 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 16 (Actual)
Dates: Start 2014-07-01 (Actual); Primary Completion 2017-03-08 (Actual); Study Completion 2018-03-08 (Actual)

PRIMARY OUTCOMES:
Concussion symptom resolution | 6 weeks
  Symptom self-reports; improvement reflected by points on the scale
Neuropsychological testing | 6 weeks
  Improved cognitive performance with the treatment, reflected in standard scores on cognitive measures.
Postural stability | 6 weeks
  Improved balance with the treatment, reflected in reductions in errors on the Balance Error Scoring System (BESS).

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Bailey, PhD, Principal Investigator — University Hospitals Cleveland Medical Center
Locations (1):
- University Hospitals Case Medical Center, Cleveland, Ohio, United States

REFERENCES:
- [Background] Centers for Disease Control and Prevention. Nonfatal traumatic brain injuries related to sports and recreation activities among persons aged </=19 years--United States, 2001-2009. MMWR Morb Mortal Wkly Rep. 2011 Oct 7;60(39):1337-42. PMID 21976115
- [Background] Gagnon I, Galli C, Friedman D, Grilli L, Iverson GL. Active rehabilitation for children who are slow to recover following sport-related concussion. Brain Inj. 2009 Nov;23(12):956-64. doi: 10.3109/02699050903373477. PMID 19831492